CLINICAL TRIAL: NCT04545658
Title: Prediction of Esophageal and Lung Toxicities After Radiation (Chemo) Therapy for Lung Cancer Management
Brief Title: Prediction of Esophageal and Lung Toxicities After Radiation (Chemo) Therapy
Acronym: PTOP-RT
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PTOP-RT (29BRC20.0154)
Record Dates: First submitted 2020-08-10; First posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
(Chemo)-radiotherapy is the gold standard therapeutic treatment for patients with locally advanced lung cancer non accessible or ineligible for surgery. While some progress occurred regarding progression free survival and overall survival thanks to recent advances (i.e., durvalumab), prediction of pulmonary and esophageal toxicity, remains insufficiently accurate. Current dose-volume histograms (DVH) do not account for spatial dose distribution and strict application of current dose constraints does not prevent toxicity events in some of the treated patients. The goal of this work was to investigate the added predictive value of the radiomics approach applied to dose maps regarding acute and late toxicity in both lungs and the esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated by (chemo)-radiotherapy for a primary lung cancer by radiotherapy

Exclusion Criteria:

* Incomplete treatment

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stage I, II, III lung cancer patients treated with (chemo)-radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Prediction of Acute Pulmonary Toxicity | Up to 6 months
  The model's performance will be evaluated based on the observed rate of Acute Pulmonary Toxicity using classification metrics (area Under the curve, balanced accuracy).
Prediction of Late Pulmonary Toxicity | Between 6 months and 2 years after radiotherapy
  The model's performance will be evaluated based on the observed rate of Late Pulmonary Toxicity using classification metrics (area Under the curve, balanced accuracy).
Prediction of Acute Oesophageal Toxicity | Up to 6 months
  The model's performance will be evaluated based on the observed rate of Acute Oesophageal Toxicity using classification metrics (area Under the curve, balanced accuracy).
Prediction of Late Oesophageal Toxicity | Between 6 months and 2 years after radiotherapy
  The model's performance will be evaluated based on the observed rate of Late Oesophageal Toxicity using classification metrics (area Under the curve, balanced accuracy).

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, Finistère, France